CLINICAL TRIAL: NCT03012581
Title: Secured Access to Nivolumab for Adult Patients With Selected Rare Cancer Types
Acronym: AcSé
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government); Ligue contre le cancer, France (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0105/1611; 2016-002257-37 (EudraCT Number)
Record Dates: First submitted 2017-01-02; First posted 2017-01-06 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma, Renal Cell; Head and Neck Neoplasm; Skin Neoplasms; Microsatellite Instability; Penile Neoplasms; Cancer With POLE Exonucleasic Domain Mutation
MeSH Terms: conditions — Carcinoma, Renal Cell; Head and Neck Neoplasms; Skin Neoplasms; Microsatellite Instability; Penile Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab 240 mg IV over 60 minutes every 14 days.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Treatment
  Other Names: Opdivo

SUMMARY:
This is a Phase 2, non-randomised, open-label, multicentric study to investigate the efficacy and safety of nivolumab monotherapy in 6 cohorts of patients with specific rare cancers who have unresectable locally advanced or metastatic disease, which is resistant or refractory to standard therapy, or for which standard therapy does not exist, or is not considered appropriate, and for which no other experimental treatment options are available.

DETAILED DESCRIPTION:
The study plans to enrol up to 300 patients in total. Eligible patients who have provided their written informed consent for study participation will be assigned to one of 6 cohorts determined by indication:

* Cohort 1: Non-clear cell RCC
* Cohort 2: Rare head and neck cancer
* Cohort 3: Rare skin cancer
* Cohort 4: non-colorectal cancers with microsatellite instability (MSI-nonCRC)
* Cohort 5: Penile cancer
* Cohort 6: POLE exonucleasic domain mutated cancer

Between 20 and 50 patients will be enrolled in each cohort, with the exception of the cohort 1 (Non-clear cell RCC) and cohort 3 (Rare skin cancer). Following the amendment 6, up to a maximum of 20 additional patients may be included in the cohort 1 (Non-clear cell RCC) or cohort 3 (Rare skin cancer), within the limit of 300 patients to be included in total, due to potential signals observed in some subsets.

The study will use a two-stage Bayesian enrichment design. The first stage treats all patients from the different cohorts with the investigational product and identifies possibly sensitive indications. The second stage will compare outcomes among subsets of patients in the identified cohorts to distinguish between subpopulations of patients who may benefit from the treatment and patients for whom there is no evidence of efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient information sheet and written informed consent form signed.
2. Histologically confirmed diagnosis of a pathology corresponding to one of the following selected cancer types:

   * Non-clear cell renal-cell carcinomas: papillary renal cell carcinoma (pRCC, type I, type II and non-classified pRCC), chromophobe RCC (ChRCC), renal medullary carcinoma (RMC), collecting duct/Bellini duct carcinoma (CDC), microphthalmia-associated transcription (MiT) family translocation renal cell carcinoma (tRCC), renal cell carcinoma with a prominent sarcomatoid component (sarcRCC).From the 51st patient included in this cohort, only the following histological type will be selected: collecting duct/Bellini duct carcinoma (CDC).
   * Rare head and neck cancers: principal and accessory salivary gland tumours, facial tissue tumours.
   * Rare skin cancers: adnexal carcinomas, basal cell carcinoma resistant to vismodegib.From the 51st patient included in this cohort, only the following histological type will be selected: Basal Cell carcinoma.
   * Non-colorectal cancers with microsatellite instability determined locally by immunohistochemistry or polymerase chain-reaction (PCR)
   * Squamous cell carcinoma of penis.
   * Any non MSI-high cancer with POLE exonucleasic domain mutation (somatic or germline) in hotspots (codons 286, 411, 424 and 459) or other germline or somatic variants with high probability of pathogenesis according to in silico assessment by the INCa ad hoc biology group.
3. Metastatic disease or unresectable locally advanced malignancy that is resistant or refractory to standard therapy or for which standard therapy does not exist or is not considered appropriate by the Investigator.
4. Aged ≥18 years old.
5. Measurable disease according to RECIST v1.1 guidelines for solid tumours.
6. Able to provide a formalin fixed/paraffin embedded (FFPE) biopsy sample of a metastatic site or primitive tumour tissue.

   Note: Patients for whom suitable archived biopsy material is not available must be willing to undergo a biopsy of a tumour lesion prior to study entry, unless this is medically contraindicated (e.g. site inaccessible or patient safety concerns).
7. Patients must have a mandatory treatment-free interval of at least 21 days following previous systemic anti-cancer treatments.
8. Patients who have received previous systemic anticancer treatment and/or radiotherapy should have recovered from any treatment related toxicity, to a level of ≤ grade 1 (according to NCI-CTCAE criteria, v 4.0) with the exception of Grade 2 alopecia.
9. Adequate hematologic function (absolute neutrophil count (ANC) ≥1.0 x10⁹/L, platelets ≥100 x10⁹/L, haemoglobin (Hb) ≥9 g/L) measured within 14 days of treatment initiation.
10. Adequate renal function (creatinine clearance ≥50 mL/min using the glomerular filtration rate (MDRD) or CKI EPI method) measured within 14 days of treatment initiation.
11. Adequate hepatic function (serum bilirubin ≤1.5 x the reference upper limit of normal (ULN) unless due to Gilbert's syndrome; aspartate aminotransferase (ASAT) and alanine aminotransferase (ALAT) ≤2.5 x ULN) measured within 14 days of treatment initiation. For patients with documented liver metastasis ASAT/ALAT ≤5 x ULN is acceptable.
12. Strictly normal blood levels of calcium and magnesium, measured within 14 days of treatment initiation.
13. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤1.
14. Estimated life expectancy ≥90 days.
15. Patients who are sexually active must agree to use a medically accepted method of contraception (e.g. implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner, for participating women; condoms for participating men) or practice complete abstinence, beginning 14 days before the first administration of investigational product (IP), while on treatment and for at least 5 months after the last administration of IP for female patients, and 7 months after the last administration of IP for male patients.
16. Women of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to the first administration of IP. If urine test results are positive or cannot be confirmed as negative, a serum pregnancy test will be required.
17. Women who are breastfeeding should discontinue nursing prior to the first administration of IP and for at least 90 days after the last administration of IP.
18. Patients must be affiliated to a Social Security System or equivalent.

Exclusion Criteria:

1. Prior treatment with an anti-PD1 or anti-PD-L1 antibody
2. Eligible, and willing, to participate in a clinical trial of an alternative anticancer therapy targeting their disease which is open to accrual in France.
3. Concurrent steroid medication at a dose greater than prednisone 10 mg/day or equivalent.
4. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
5. History of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
6. History of severe hypersensitivity reaction to any monoclonal antibody therapy
7. Radiotherapy (except for brain and extremities) within 21 days prior to the first administration of IP.
8. Treatment with other investigational drugs or participation in another clinical trial within 21 days prior to the first administration of IP or concomitantly with the trial.
9. Has known symptomatic central nervous system (CNS) metastases. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
10. Has known carcinomatous meningitis or a history of leptomeningeal disease.
11. Serum creatinine >1.5 x ULN or glomerular filtration rate (GFR) <50 mL/min.
12. Other malignancies within the past 5 years other than basal cell skin cancer or carcinoma in situ of the cervix.
13. Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy.
14. Active or chronic hepatitis B, hepatitis C and/or human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies), or a known history of active Tuberculosis bacillus.
15. Has received a live vaccine within 30 days of planned start of study treatment. Note: Seasonal influenza vaccines for injection are generally inactivated vaccines and are allowed.
16. Active alcohol or drug abuse.
17. Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule.
18. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate | measured at the first scheduled disease assessment following study treatment initiation (Day 84, ± 7 days)
  ORR will be assessed per cohort by an IRC according to RECIST v1.1.

SECONDARY OUTCOMES:
Progression-free survival | From date of inclusion until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 36 months
  Assessed according to RECIST v1.1
Overall survival | From date of inclusion until the date of death from any cause, assessed up to 36 months
Best response | From inclusion up to 36 months
  Assessed according to RECIST v1.1
Response duration | from first observation of objective response until date of first documented progression or date of death from any cause, whichever comes first, assessed up to 36 months
  Assessed according to RECIST v1.1
Time to response | from inclusion first observation of objective response, assessed up to 36 months
  Assessed according to RECIST v1.1
Frequency and severity of adverse events | from inclusion until 100 days after last dose of investigational product
  assessed according to the NCI-CTCAE v4
Objective response rate in subgroups of subjects with high versus low expression (cutoff set at the median for the population measured) of different immune markers (PD-L1, CD4+, FOXP3+, Fas-L, OX40, VEGF, CD31; CD34) | measured at the first scheduled disease assessment following study treatment initiation (Day 84, ± 7 days)
  ORR will be assessed per cohort by an IRC according to RECIST v1.1.
Progression-free survival in subgroups of subjects with high versus low expression (cutoff set at the median for the population measured) of different immune markers (PD-L1, CD4+, FOXP3+, Fas-L, OX40, VEGF, CD31; CD34) | From date of inclusion until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 36 months
  Assessed according to RECIST v1.1.
Overall survival in subgroups of subjects with high versus low expression (cutoff set at the median for the population measured) of different immune markers (PD-L1, CD4+, FOXP3+, Fas-L, OX40, VEGF, CD31; CD34) | From date of inclusion until the date of death from any cause, assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien Marabelle, MD, Principal Investigator — Gustave Roussy Cancer Campus
Locations (1):
- Gustave Roussy Cancer Campus, Villejuif, France

IPD SHARING:
Plan to Share IPD: No